CLINICAL TRIAL: NCT05238051
Title: The Role of Gastric Residual Volume Measurement in Achieving Target Calories in the Intensive Care Unit: A Randomized Controlled Study
Brief Title: Gastric Residual Volume Measurement in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, Alparslan Koc, Principal Investigator, Erzincan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRVROLE
Record Dates: First submitted 2022-01-21; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Preventing Malnutrition
Keywords: gastric residual volume; malnutrition; target calorie; intensive care unit; enteral nutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Gastric residual volume (GRV) was measured in one group and not in the other. Nutrition was started at an infusion rate of 20 ml/hour in the GRV group. The GRV was measured every four hours. When it was less than 200 ml, the infusion rate was increased by 20 ml/hour. The infusion rate, which was increased every four hours according to the GRV, was continued constantly when the target calorie was reached. It was kept constant when the GRV was above 200 ml, and then the feeding rate was reduced to half when the GRV volume was above 400 ml. In four patients, enteral nutrition was discontinued due to melena and excluded from the study. In six patients with persistently high GRV values, enteral nutrition was discontinued and parenteral nutrition initiated. The study was completed with 62 patients. GRV (n=31) and Non-GRV (n=31).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric residual volume group (No Intervention): Patients undergoing enteral nutrition with continuous infusion and intermittent gastric residual volume measurement in the intensive care unit
- Non- Gastric residual volume group (Experimental): Patients undergoing enteral nutrition with continuous infusion and intermittent gastric residual volume measurement was not measured in the intensive care unit
  Interventions: Other: Gastric residual volume measurement stopped.

INTERVENTIONS:
Other: Gastric residual volume measurement stopped. — GRV is checked during routine enteral nutrition, but we think that GRV prolongs the time to reach target calories and does not reduce complications.
  Arms: Non- Gastric residual volume group

SUMMARY:
Nutritional support is considered a key component of the treatment strategy for intensive care patients. Malnutrition, energy protein, and inadequate or excessive intake of other nutrients have measurable effects on tissues, body structure, body function, and clinical outcomes of patients receiving treatment. It increases hospital-acquired infections, hospitalizations, and intensive care prolongs and leads to complications. This study aimed to observe the time to reach target calories, nutritional failures, and complications during feeding in measured and unmeasured gastric residual volume patients receiving enteral nutrition under ventilation in the intensive care unite.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilatory support
* open enteral route (nasogastric/PEG)

Exclusion Criteria:

* History of gastrointestinal bleeding,
* parenteral nutrition support,
* hospital stay of fewer than two days,
* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
The difference in the time to reach target calories in patients with gastric residual volume measurement compared to those without gastric residual volume measurement. | 10 days
  The difference in the time to reach target calories in patients with gastric residual volume measurement compared to those without gastric residual volume measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Binali Yildirim university, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marik PE. Enteral nutrition in the critically ill: myths and misconceptions. Crit Care Med. 2014 Apr;42(4):962-9. doi: 10.1097/CCM.0000000000000051. PMID 24296860
- [Background] Elke G, Felbinger TW, Heyland DK. Gastric residual volume in critically ill patients: a dead marker or still alive? Nutr Clin Pract. 2015 Feb;30(1):59-71. doi: 10.1177/0884533614562841. Epub 2014 Dec 18. PMID 25524884